CLINICAL TRIAL: NCT06795360
Title: Weight Changes After Incretin-mimetics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Lisa Morselli, MD PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00052666
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; weight loss; weight gain
MeSH Terms: conditions — Obesity; Weight Loss; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- incretin mimetic discontinuation (Experimental): This study will enroll people who are taking an injectable weight loss drug, have lost weight with the help of this drug, and are required by their health insurance plan to discontinue treatment. They will be studied right before their medication runs out, and 3 months later
  Interventions: Other: discontinuation of weight loss medication

INTERVENTIONS:
Other: discontinuation of weight loss medication — Participants will be studied right before their injectable weight loss medication runs out, and 3 months later

SUMMARY:
The goal of this study is to identify people at risk of weight regain after stopping an injectable weight loss drug. The main question the investigators aim to answer is: Can weight regain be predicted by measuring circulating Agouti-related peptide, a small protein coming from the brain?

DETAILED DESCRIPTION:
This study will enroll people who are taking an injectable weight loss drug, have lost weight with the help of this drug, and are required by their health insurance plan to discontinue treatment. Participants will first be screened for health conditions that would prevent them from entering the study. Once enrolled, participants will be asked to have the following testing while still on the injectable weight loss drug: body weight measurement, body composition (fat and lean mass), resting energy expenditure (calories burned), multiple blood draws after overnight fast and after drinking and nutritional shake urine collection, urine collection, measurement of heart rate, measurement of physical activity and sleep, questionnaires. Participants will then stop taking the injectable weight loss drug when the prescription runs out, and the same tests will be repeated 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years or older
* men and women
* prescribed an incretin-mimetic for weight loss and for whom insurance coverage for this specific drug will lapse
* any ethnicity

Exclusion Criteria:

* weight > or = 400 lb
* type 1 or type 2 diabetes
* patients taking steroid medications
* anemia
* heart disease
* advanced kidney disease (CKD stage 4 and 5)
* decompensated liver disease
* hyperthyroidism
* untreated hypothyroidism
* active cancer
* post solid organ or bone marrow transplant
* HIV/AIDS
* pregnancy/plan for pregnancy in the next 6 months
* breastfeeding
* post-menopausal women
* current smoker
* current recreational drug use
* night shift or rotating shift workers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2031-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
weight change | 3 months
  weight trajectories in the 3 months after treatment discontinuation
fasting and post-prandial circulating AgRP | 3 months
  Circulating AgRP will be measured after an overnight fast and during a 3-hour mixed meal test, at baseline (while still on injectable weight loss drug) and 3 months later. The mixed meal will consist in a nutrtional shake consumed in 5 min.

SECONDARY OUTCOMES:
subjective hunger ratings | 3 months
  Participants will be asked to rate current hunger with a visual analogue scale in fasting conditions and hourly during a 3-hour mixed meal test. This will be done at baseline (while still on injectable weight loss drug) and 3 months after treatment discontinuation. Scores go from 0 to 100, with 0 indicating "Not hungry at all" and 100 indicating "Extremely hungry".
resting metabolic rate (RMR) | 3 months
  RMR will be measured in fasting conditions at baseline (while still on injectable weight loss drug) and 3 months after treatment discontinuation.
RMR adaptation | 3 months
  RMR adaptation will be estimated baseline (while still on injectable weight loss drug) and 3 months after treatment discontinuation. RMR adaptation will be defined as the difference between measured and predicted RMR. Predicted RMR will be computed with a linear regression equation obtained from baseline data from the whole cohort.
body composition | 3 months
  Body composition (fat mass, fat-free mass) will be measured at baseline and 3 months later by DXA

IPD SHARING:
Plan to Share IPD: Yes
All datasets that pass quality control procedures and any other data that are deemed necessary to validate and replicate research findings will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: The data deposited will be made available to all investigators in the research community as soon as possible but no later than 12 months from the completion of the funding period or upon acceptance of the data for publication and release from journals, whichever is earlier. Requests for data will be filled in a timely manner, usually within 2 to 6 weeks of the request, depending on the chronological position of the request within the queue. In addition, research data which documents, supports, or validates the published research findings, will be made available (electronically or mailed hard-copies) upon request to NIH-funded research programs. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: Other researchers will be able to access the IPD if they submit a proposal that describes planned analyses. A data sharing agreement must be signed. Researchers interested in the IPD can contact Dr. Morselli by email and send documents by email. Dr. Morselli will then share the ICR.